CLINICAL TRIAL: NCT01470235
Title: Hypodontia and Ovarian Cancer - the Connection Between Dental Agenesis and Epithelial Cancers, Especially Ovarian Cancer.
Brief Title: Hypodontia and Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cancer Society (Other); Arvid-Nilsson Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: Hypodontovariancancer2011
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Ovarian Cancer; Hypodontia; Breast Cancer; Colon Cancer
Keywords: screening; genetic; cancer
MeSH Terms: conditions — Ovarian Neoplasms; Anodontia; Breast Neoplasms; Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 5ml EDTA full blood for DNA analysis.
  1 PAX-tube for RNA analysis. Biopsi from removed tumor-tissue for DNA analysis. Both preserved in Danish Cancer Biobank for later analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Ovarian Cancer: Women treated for ovarian cancer at the departments of obstetrics and gynecology, Aarhus University Hospital and Rigshospitalet, Copenhagen.
  Expected recruitment: 200
- Control patients: Women referred to the departments of obstetrics and gynecology in Aarhus University Hospital and Rigshospitalet, Copenhagen on benign indication.
  Expected recruitment: 200.
- HBOC/HNPCC: Patients registered in the large Danish Register of HBOC( hereditary breast and ovarian cancer) and HNPCC (hereditary nonpolyposis colorectal cancer).
  Expected recruitment: 200.

SUMMARY:
The purpose of this project is to examine whether the risk of developing ovarian cancer is increased in Danish women with congenital missing teeth as a result of their failure to develop (hypodontia). Should this prove to be the case, these women could be offered regular clinical controls and prophylactic removal of their ovaries when menopause enters and the ovaries are no longer functional (producing hormones).

If there is a connection between congenital hypodontia and the development of different types of cancer, the investigators will perform a genetic screening in families with increased risk of cancer and hypodontia for changes in relevant genes, based on the current literature. The investigators hereby search for new genes, which in a changed form leads to an increased risk of cancer and thereby enables us to perform genetic screening in risk families.

ELIGIBILITY:
Inclusion Criteria:

* confirmed suspicion of ovarian cancer.

Exclusion Criteria:

* suspicion of ovarian cancer disproved.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women referred to the department of obstetrics/gynecology under the diagnosis ovarian cancer obs. pro.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence rates of hypodontia in women with ovarian cancer | one year

SECONDARY OUTCOMES:
Genetic causes for hypodontia and ovarian cancer | two years
Prevalence rates of hypodontia in patients with a known risk for epithelial cancer | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jan Blaakaer, Professor, MD, DMSc, Study Director — Aarhus University Hospital; Maria Cathrine C. V. Schmidt, MD, Ph.d.-student, Principal Investigator — Aarhus University Hospital; Charlotte Soegaard, MD, ph.d., Study Chair — Aarhus University Hospital; Lone Sunde, Associate Professor, PhD, Study Chair — Aarhus University Hospital; Claus Hoegdall, Professor, Study Chair — Copenhagen University Hospital at Herlev; Michala O. Lexner, Dentist, PhD, Study Chair
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Skejby, Aarhus
  - Copenhagen University Hospital, Copenhagen Ø, Copenhagen

REFERENCES:
- [Background] Chalothorn LA, Beeman CS, Ebersole JL, Kluemper GT, Hicks EP, Kryscio RJ, DeSimone CP, Modesitt SC. Hypodontia as a risk marker for epithelial ovarian cancer: a case-controlled study. J Am Dent Assoc. 2008 Feb;139(2):163-9. doi: 10.14219/jada.archive.2008.0132. PMID 18245684
- [Background] Eisinger F, Burke W, Sobol H. Management of women at high genetic risk of ovarian cancer. Lancet. 1999 Nov 6;354(9190):1648. doi: 10.1016/S0140-6736(05)77137-3. No abstract available. PMID 10560705
- [Background] Cobourne MT. Familial human hypodontia--is it all in the genes? Br Dent J. 2007 Aug 25;203(4):203-8. doi: 10.1038/bdj.2007.732. PMID 17721480
- [Background] Rolling S. Hypodontia of permanent teeth in Danish schoolchildren. Scand J Dent Res. 1980 Oct;88(5):365-9. doi: 10.1111/j.1600-0722.1980.tb01240.x. PMID 6936762
- [Background] Rolling S, Poulsen S. Oligodontia in Danish schoolchildren. Acta Odontol Scand. 2001 Apr;59(2):111-2. doi: 10.1080/000163501750157298. PMID 11370748
- [Background] Marchini S, Marabese M, Marrazzo E, Mariani P, Cattaneo D, Fossati R, Compagnoni A, Fruscio R, Lissoni AA, Broggini M. DeltaNp63 expression is associated with poor survival in ovarian cancer. Ann Oncol. 2008 Mar;19(3):501-7. doi: 10.1093/annonc/mdm519. Epub 2007 Nov 12. PMID 17998283
- [Background] Lammi L, Arte S, Somer M, Jarvinen H, Lahermo P, Thesleff I, Pirinen S, Nieminen P. Mutations in AXIN2 cause familial tooth agenesis and predispose to colorectal cancer. Am J Hum Genet. 2004 May;74(5):1043-50. doi: 10.1086/386293. Epub 2004 Mar 23. PMID 15042511